CLINICAL TRIAL: NCT02374463
Title: Improving Balance and Mobility in Older Veterans
Brief Title: Improving Balance and Mobility
Acronym: MMBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E1574-P; 1I21RX001574-01A1 (NIH); NCT02234817 (obsolete NCT alias)
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Postural Balance; Accidental Falls; Mobility Limitation
Keywords: Balance; Fall Risk; Older Adults; Tai Chi; Multimodal Balance Intervention
MeSH Terms: conditions — Mobility Limitation | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodality Balance Intervention (MMBI) (Experimental): Multimodality Balance Intervention (MMBI)
  Interventions: Behavioral: MMBI
- Tai Chi (Active Comparator): Tai Chi Intervention
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: MMBI — Multimodality Balance Intervention (MMBI): Our MMBI will be held 3-times a week for an hour and will consist of a group dynamic balance class (30 minutes), a supervised obstacle course (10 minutes), and lower extremity and core strengthening (20 minutes). The group exercise classes will focus on dynamic weight shifts with an emphasis on the lateral and diagonal directions. Over the 6 months of class, the exercises will gradually increase in difficulty to challenge balance. A skilled instructor will lead each class and 1-2 assistants will be present to assist with fall risk prevention. The supervised obstacle course will focus on obstacle negotiation, gait over challenging surfaces, and moving in lateral, diagonal, and backward directions. Finally, strength training of the lower extremities and core will focus on strengthening major muscles of the lower extremity and core utilizing commonly available gym equipment, ankle weights and body weight.
  Arms: Multimodality Balance Intervention (MMBI)
Behavioral: Tai Chi — Tai Chi Intervention: The supervised Tai Chi class will be held 3-times a week for one hour. All Tai Chi classes will be taught in a group setting by an experienced instructor. The emphasis during the class will be on standing movements, body alignment, weight shift and changes of direction. Movements will be adapted as the class progresses to increase the difficulty of weight shift and change in direction over time so that participants balance is continually challenged throughout the 6 months. Chairs or hand rails will be available for the participants to use as needed for balance recovery.
  Arms: Tai Chi

SUMMARY:
Falls are dangerous leading to injuries and even death. The VA has made fall prevention a priority, but effective programs only reduce falls by 30%. Tai Chi, a standing exercise program, has been effective at improving balance but may not prevent falls. Most falls occur during walking when an individual experiences a slip or a trip. Programs that focus on walking, stepping, and recovery from a slip may be more effective at fall reduction. This study will compare Tai Chi to a novel multimodal balance intervention (MMBI). MMBI focuses on standing balance, walking, stepping, strength training, and recovery from a slip. The Investigators believe that the MMBI program will be more effective than Tai Chi at improving balance and preventing falls in older Veterans and the Investigators will use the results of this study to develop a larger study on fall prevention in older Veterans.

DETAILED DESCRIPTION:
Background: Falls are currently the leading cause of injurious death and non-fatal injuries for adults over the age of 65. Older Veterans may be at greater risk for falls due to their high burden of medical co-morbidity. The VA has made research into fall prevention a high priority. Falls are complex with numerous deficits including impaired balance, decreased postural control, muscle weakness, and an inability to successfully negotiate environmental hazards. Tai Chi is currently considered to be one of the most effective fall prevention exercise interventions, with an endorsement from the Centers for Disease Control and Prevention (CDC) which widely influences health care policy. However, there are few studies comparing Tai Chi with another active intervention. Tai Chi may generally improve balance, decrease fall risk, and provides a general lower body strengthening. However, Tai Chi may not sufficiently improve gait and dynamic mobility and does little to target obstacle negotiation, one of the largest contributors to a fall. The majority of falls occur during walking, with slips and trips being the most common causes and targeted interventions focused on improving stepping and walking ability may be even more effective at improving balance and reducing falls.

The Investigators plan to enroll 56 older (age > 65 years) community dwelling Veterans with a history of a fall in the last year who are at high risk for a recurrent fall. After baseline testing participants will be randomized to either MMBI or a Tai Chi intervention modeled after the Tai Chi Moving for Better Balance Program. All participants will participate in a group exercise class in their assigned intervention for 1 hour, 3 times per week for 24 weeks. After the completion of 24 weeks of exercise group changes will be compared for 1) balance (4-square step test); 2) mobility and fall risk (functional gait assessment); 3) rate of falls; 4) lower extremity isometric strength testing (biodex); and 5) body composition. The investigators also plan for follow all participants for 6 months after completion of the intervention to examine differences in fall rates after the cessation of the program between the groups.

Impact: This research directly benefits Veterans as it may lead to new and effective interventions that could reduce fall risk, injury-related hospitalization and death in older Veterans. MMBI is also readily exportable to the community and with minimal resources could be widely implemented at other VAs as part of standard of care, similar to Managing Overweight and/or Obesity for Veterans Everywhere! (MOVE!). Results from this SPIRE grant will be used to power a larger randomized clinical trial that will examine the effectiveness of the two interventions to reduce rate of falls and risk of falling in older Veterans at high risk for falls.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* Mobility and balance limitations as demonstrated by a self-reported fall within the past year or requiring greater than 8 seconds to complete the 4-square step test

Exclusion Criteria:

* Cardiovascular Risks: Poorly controlled hypertension (>160/100); Class III or IV congestive heart failure (CHF); or patient report of: symptomatic angina at rest or during exercise, syncope without known resolution of cause, or a significant coronary event (such as a MI) in the past six months
* Chronic obstructive pulmonary disease (COPD) requiring home oxygen
* Contraindications to resistance training, including a self-reported history of intracranial or retinal bleeding in the last year or Diabetes with active proliferative retinopathy
* Patient report of significant spinal stenosis that would limit participation in the exercise intervention -Dementia (on medical record review or mini-mental status exam score <24).
* Non-ambulatory mobility status or a transtibial or transfemoral amputation
* Other severe medical illness or condition that would preclude safe participation in the study as determined by the study team

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Ira Katzel, MD PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- See also: Exercise and Physical Fitness — http://www.nlm.nih.gov/medlineplus/exerciseandphysicalfitness.html
- See also: Falls — http://www.nlm.nih.gov/medlineplus/falls.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Older community dwelling veterans (age > 65 years) with evidence of balance dysfunction (Four Square Step Test > 8 seconds) and or history of falling were recruited for this study. 41 subjects signed informed consent. 10 subjects were ineligible, 4 dropped out prior to completing baseline testing resulting in 27 subjects who were randomized.
Groups:
- MMBI: Multimodality Balance Intervention (MMBI): The Investigator's MMBI class will be held 3-times a week for an hour and will consist of a group dynamic balance class (30 minutes), a supervised obstacle course (10 minutes), and lower extremity and core strengthening (20 minutes). The group exercise classes will focus on dynamic weight shifts with an emphasis on the lateral and diagonal directions. Over the 6 months of class, the exercises will gradually increase in difficulty to challenge balance. A skilled instructor will lead each class and 1-2 assistants will be present to assist with fall risk prevention. The supervised obstacle course will focus on obstacle negotiation, gait over challenging surfaces, and moving in lateral, diagonal, and backward directions. Finally, strength training of the lower extremities and core will focus on strengthening major muscles of the lower extremity and core utilizing commonly available gym equipment, ankle weights and body weight.
Period: Overall Study
Arm/Group | MMBI | Tai Chi
Started | 15 | 12
Completed | 12 | 9
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- MMBI: Multimodality Balance Intervention (MMBI)
- Total: Total of all reporting groups
Arm/Group | MMBI | Tai Chi | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (8.2) | 75.7 (5.1) | 75.1 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27
four square step test [Mean (Standard Deviation); unit: seconds] — For this test, subjects step over a grid of canes laid out in a square pattern on the floor. Higher values in seconds are associated with increased fall risk.
  seconds | 11.6 (2.0) | 12.3 (3.4) | 12 (3)
% body fat [Mean (Standard Deviation); unit: % body fat] | 37.7 (8.9) | 38.8 (5.0) | 38.2 (4.1)
isometric strength hip [Mean (Standard Deviation); unit: newton squared] — isometric strength R hip measured using biodex
  newton squared | 46.2 (17.2) | 48.5 (28.1) | 47.1 (22.3)
isometric strength knee [Mean (Standard Deviation); unit: newton squared] — isometric strength R knee measured using biodex
  newton squared | 114.6 (49.8) | 127.4 (31.1) | 120.2 (27.2)

OUTCOME MEASURES:

1. Primary Outcome: Balance and Lateral Mobility Assessed by the Four Square Step Test
Description: the Four Square Step Test assesses dynamic balance and coordination through stepping forwards, sideways, and backwards in a timed fashion. The four square step test is timed in seconds. Higher scores are associated with worse outcome. Individuals with higher scores are at increased risk of falling with some using a score of 15 seconds or higher as being at high risk for falls. The minimum value one would see in young healthy populations for this test is 5 seconds. The maximum value is 60 seconds. If they are deemed unable to complete the value is not reported
Time Frame: The FSST was assessed at 6 month (post) and at baseline (pre)
Population: the change in four square step test score is calculated as the 6 month (post) - the baseline value (pre)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MMBI | Tai Chi
Number analyzed (Participants) | 12 | 9
seconds | -1.8 (0.9) | -0.6 (0.3)
Statistical Analysis 1: Comparison: MMBI vs Tai Chi; within group change was assessed; Test type: Superiority; p < 0.05, t-test, 2 sided — P value not adjusted for multiple comparisons

2. Secondary Outcome: Functional Gait Analysis
Description: The Functional Gait Assessment (FGA) is designed to assess postural stability during gait. The measure is calculated by summing the scores for 10 gait related tasks. Each task is scored from 3 to 0, where 3 is the best possible performance (normal) and 0 indicates severe impairment related to the task. The best possible score is 30 and the worst possible score is 0. Higher values are associated with better outcome. A value of 22/30 and below is associated with high risk of falling in the community.
Time Frame: FGA ws measured at 6 months (post) and at baseline (pre)
Population: The change in FGA was calculated as the value at 6 months (post)- the value at baseline (pre)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMBI | Tai Chi
Number analyzed (Participants) | 12 | 9
score on a scale | 7.28 (3.64) | -0.5 (0.3)
Statistical Analysis 1: Comparison: MMBI vs Tai Chi; Test type: Superiority; p = 0.08, ANOVA — p value not adjusted for multiple comparisons

3. Secondary Outcome: Change in Strength R Knee Biodex
Description: Change in isometric strength R knee assessed using the biodex measured before and after intervention. Change was calculated as value at 6 months (post)-value at baseline (pre).Higher values are a better outcome
Time Frame: Strength at the R knee was assessed at 6 months (post) and at baseline (pre)
Measure: Mean (Standard Deviation); unit: newton squared
Arm/Group | MMBI | Tai Chi
Number analyzed (Participants) | 12 | 9
newton squared | 21.8 (10.5) | -16.2 (8.1)
Statistical Analysis 1: Comparison: MMBI vs Tai Chi; Test type: Superiority; p = 0.6, ANOVA; not adjusted for multiple comparisons

4. Secondary Outcome: Number of Subjects Who Reported Falls
Description: This is the number of subjects who self-reported at least one fall, and does not include trips or near falls. This measure does not include the total number of falls as there were several participants who reported more than one fall.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- MMBI: Multimodality Balance Intervention (MMBI):
Arm/Group | MMBI | Tai Chi
Number analyzed (Participants) | 15 | 12
participants | 3 | 3
Statistical Analysis 1: Comparison: MMBI vs Tai Chi; Test type: Superiority; p = 0.84, Chi-squared — Not adjusted for multiple comparisons; exploratory aim prespecified
Statistical Analysis 2: Comparison: MMBI vs Tai Chi; Test type: Superiority; p = 0.4, Chi-squared

5. Secondary Outcome: Change in Strength R Hip Using Biodex
Description: Assessment of change in strength using biodex. Higher values are associated with better outcome
Time Frame: Strength in the R hip was assessed at 6 months (post) and at baseline (pre)
Population: Change calculated as 6 month value (post)- baseline value (pre)
Measure: Mean (Standard Deviation); unit: newton squared
Arm/Group | MMBI | Tai Chi
Number analyzed (Participants) | 12 | 9
newton squared | 10.4 (5.2) | -10.1 (5.1)
Statistical Analysis 1: Comparison: MMBI; Test type: Superiority; p = 0.3, ANOVA — not adjusted for multiple comparisons

6. Other Pre Specified Outcome: Percent Body Fat
Description: change in total body fat measured using Dual-energy X-ray absorptiometry (DXA). Value was calculated as value at 6 months (post) - value at baseline (pre)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | MMBI | Tai Chi
Number analyzed (Participants) | 12 | 9
percentage of body fat | -0.37 (0.19) | -0.1 (0.05)
Statistical Analysis 1: Comparison: MMBI vs Tai Chi; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Description: Prospective monitoring
Arm/Group | MMBI | Tai Chi
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/12
Other Adverse Events (participants affected / at risk) | 3/15 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMBI (N=15) | Tai Chi (N=12)
hospitalization (Gastrointestinal disorders) | 1 (1) | 1 (1) — surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMBI (N=15) | Tai Chi (N=12)
fall (Musculoskeletal and connective tissue disorders) | 3 (15) | 3 (12)

LIMITATIONS AND CAVEATS:
Interpretation of the results is limited by the modest sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT02374463/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT02374463/ICF_001.pdf